CLINICAL TRIAL: NCT06238297
Title: Rapid De-escalation of Anti-MRSA Therapy Guided by S. Aureus Nares Screening in Case of Pneumonia (SNAP Study)
Brief Title: Rapid De-escalation of Anti-MRSA Therapy Guided by S. Aureus Nares Screening in Case of Pneumonia
Acronym: SNAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Francesco Vladimiro Segala, Principal investigator, University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNAPv1.2
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pneumonia, Bacterial
Keywords: MRSA; Antimicrobial stewardship; Randomized trial; Pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients included into the intervention arm will undergo a nasal swab for MRSA and empirical anti-MRSA therapy will be discontinued f the nasal swab result is negative.
  Interventions: Diagnostic Test: MRSA nasal swab based de-escalation
- Control (No Intervention): Patients randomized into the control arm will continue pneumonia treatment as per standard of care

INTERVENTIONS:
Diagnostic Test: MRSA nasal swab based de-escalation — Patients included into the intervention arm will undergo a nasal swab for MRSA and empirical anti-MRSA therapy will be discontinued f the nasal swab result is negative.
  Arms: Intervention

SUMMARY:
The current IDSA/ATS guidelines recommend Linezolid and Vancomycin for MRSA coverage in hospitalized patients with pneumonia, which is common clinical practice in Italy. However, a nasal PCR-assay for MRSA has a high negative predictive value and can facilitate rapid antibiotic de-escalation, thereby avoiding unnecessary anti-MRSA treatments. The indiscriminate use of these drugs has contributed to the emergence of resistant S. aureus strains and has led to significant adverse effects, without providing any survival benefits. Additionally, it has increased hospital stays and associated costs. The proposed study aims to use this diagnostic tool to shorten empirical anti-MRSA treatment duration in pneumonia patients, focusing on reducing antimicrobial therapy days while measuring in-hospital mortality, length of stay and adverse drug event incidence.

DETAILED DESCRIPTION:
BACKGROUND On the basis of current IDSA/ATS guidelines antimicrobial agents such as Linezolid and Vancomycin are commonly used in hospitalized patients as an empirical treatment in community acquired pneumonias (CAPs) particularly in hospital-acquired pneumonias (HAPs) and ventilator associated pneumonias (VAPs), suggesting the empiric use of such anti-MRSA agents for patients with specific risk factors (e.g. recent hospitalization, exposure to parenteral antibiotics and/or previous isolation of these organisms, in particular from the respiratory tract) while obtaining culture data.

According to the 2023 annual report of the European Antibiotic Resistance Surveillance System (EARSS) there is a high prevalence of MRSA throughout the European territory, however, even in countries with high endemicity, the presence of MRSA has remained stable in the last years. In Italy, according to the National Antibiotic-Resistance Surveillance System AR-ISS, in 2021 the percentage of blood isolates MRSA isolates showed a reduction (29.9%) in the national territory, standing, however, at 33.6% in the Puglia region, a percentage higher than the European.

In patients with pneumonia, the nasal PCR-assay for MRSA has a high negative predictive value (NPV), with the crucial implication that a negative result can be used to guide the antibiotic de-escalation, avoiding an improper empiric use of the anti-MRSA therapy. Data supporting the clinical validity of the use of the nasal swab for MRSA as a diagnostic tool for pneumonia are robust, in this regard, as stated by the IDSA/ATS guidelines and supported by numerous retrospective studies, anti-MRSA treatment can be avoided in case of negative result, especially in non-severe CAP, thus preventing the misuse of anti-MRSA drugs.

The indiscriminate use of these drugs over time has considerably led to the selection of resistant strains of S. aureus such as Vancomycin-intermediate Staphylococcus aureus (VISA), heterogeneous VISA (hVISA) and Vancomycin-resistant Staphylococcus aureus (VRSA). Furthermore, the high risk of adverse events given by the empirical use of anti-MRSA drugs should also be noted including, among others, nephrotoxicity and ototoxicity with vancomycin and bone marrow suppression and peripheral neuropathy with linezolid, without a gain in terms of survival and with longer hospitalization stays.

In addition, the systematic use of such drugs is associated with an increase in hospital costs, where the PCR assay for MRSA has a relevant role. According to a study conducted by the Stanford University in 2021, enabling antibiotic de-escalation within 24h, its use has of facts led to a cost saving of vancomycin of $40.33 per patient.

On these assumptions, it is clear that using the nasal swab for MRSA in pneumonia diagnosis avoids the use of expensive drugs giving a large impact on health costs, while also reducing the risk of iatrogenic toxicity, hospital stay days and the duration of ventilation in VAPs.

The aim of our study is to implement the use of the nasal swab for MRSA as a diagnostic tool reducing the duration of the empirical anti-MRSA treatment in the population of hospitalized patients with pneumonia.

METHODS AND PROCEDURES. This will be a prospective, randomized single-center controlled study conducted in the Azienda Consorziale Policlinico di Bari.

The minimum sample size is 38 patients per group, for a total of 76 subjects, calculated assuming a standard deviation of 10, a power of 90% and a type I error of 5%.

The study will involve two phases: a first phase of enrollment of the subjects, with the collection of informed consent, of the anamnestic and personal data, a phase of randomization with consequent execution, within 48h from the start of the anti-MRSA empirical therapy, of the nasal swab for MRSA in the experimental group of patients. In a second step, the research assistants will continue the follow-up of the subject with cessation of the empiric treatment in case of negative result of the swab.

The implementation of these steps will be ensured by the performance of the tasks foreseen for each unit. Each clinical unit will:

* Enroll patients and collect demographic, clinical, and biochemical data at baseline, as well as ensure their management according to guidelines and scientific evidence for the entire duration of the follow-up;
* Perform a nasal swab for MRSA in patients in the experimental group and discontinue the empirical anti-MRSA therapy if the nasal swab result is negative.
* For both arms, follow-up visits will be on day 2, 5, 7, 14, and 28 relative to the enrollment visit (day 0). At the control visits, data will be collected on the clinical course of pneumonia and laboratory tests. After discharge, the visit can also be conducted by telephone.

For more precision, eligibility criteria and primary and secondary outcomes descriptions are fully detailed in the corresponding sections.

TIMELINE The research project will have a duration of 12 months following the approval of the Ethics Committee of the University of BarI.

STATISTICAL ANALYSIS The sample size is estimated based on the main outcome measure (duration of antibiotic intake), which the investigators assume to have an average of 10 days in the control group and 2 days in the experimental group. Assuming a standard deviation of 10, a power of 90%, and a type I error of 5%, it is necessary to enroll a minimum of 34 patients per group (thus a total of 68 patients) in order to demonstrate a reduction from 10 to 2 days in the duration of antibiotic intake. To this is added an estimated 10% of cases lost to follow-up, resulting in a final sample size of 76 patients.

The statistical analysis will be conducted according to the intention-to-treat approach. In case of contamination between the two treatment groups (which is considered unlikely in this case), an analysis per protocol will also be performed and the conclusions of the study will take into account the results of both. Numerical data will be summarized as mean and standard deviation, while categorical data as absolute and relative frequency. The two groups will be compared with the Student's t-test (numerical data) and with the Chi-Square test or Fisher's test (categorical data). The effects will be expressed as mean difference or relative risk, accompanied by a 95% confidence interval. All tests will be two-tailed, and a p-value lower than 0.05 will be considered significant. The statistical analysis will be carried out with R software version 4.3 (R Foundation for Statistical Computing, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older.
* Patients hospitalized at the Azienda Consorziale Policlinico di Bari;
* Clinical diagnosis of CAP/HAP/VAP;
* Commitment by the prescribing physician to set an anti-MRSA antibiotic therapy in empirical
* Enrollement within 48h from the beginning of the empirical anti-MRSA therapy.

Exclusion Criteria:

* Febrile neutropenia or severe immunodeficiency;
* Chronic airway infection (eg cystic fibrosis);
* Suspect of extrapulmonary infection by MRSA
* Refusal by the patient or legal guardian;
* Refusal by the physician in charge of the patient to perform antibiotic de-escalation based on the result of the nasal swab;
* Enrollment after 48 hours from the beginning of the empirical anti-MRSA therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-06-03 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of antibiotic intake | From day zero to day 28

SECONDARY OUTCOMES:
In-hospital mortality | From day zero to day 28
Hospital lenght-of stay | From day zero to day 28 or until discharge
Incidence of severe pneumonia requiring mechanical ventilation | From day zero to day 28 or until discharge
Incidence of drug-related adverse outcomes | From day zero to day 28
Hospital costs | From day zero to day 28 or until discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Bari "Aldo Moro", Bari, Italy

REFERENCES:
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Dangerfield B, Chung A, Webb B, Seville MT. Predictive value of methicillin-resistant Staphylococcus aureus (MRSA) nasal swab PCR assay for MRSA pneumonia. Antimicrob Agents Chemother. 2014;58(2):859-64. doi: 10.1128/AAC.01805-13. Epub 2013 Nov 25. PMID 24277023
- [Background] Parente DM, Cunha CB, Mylonakis E, Timbrook TT. The Clinical Utility of Methicillin-Resistant Staphylococcus aureus (MRSA) Nasal Screening to Rule Out MRSA Pneumonia: A Diagnostic Meta-analysis With Antimicrobial Stewardship Implications. Clin Infect Dis. 2018 Jun 18;67(1):1-7. doi: 10.1093/cid/ciy024. PMID 29340593
- [Background] Mergenhagen KA, Starr KE, Wattengel BA, Lesse AJ, Sumon Z, Sellick JA. Determining the Utility of Methicillin-Resistant Staphylococcus aureus Nares Screening in Antimicrobial Stewardship. Clin Infect Dis. 2020 Aug 22;71(5):1142-1148. doi: 10.1093/cid/ciz974. PMID 31573026
- [Background] Dadgostar P. Antimicrobial Resistance: Implications and Costs. Infect Drug Resist. 2019 Dec 20;12:3903-3910. doi: 10.2147/IDR.S234610. eCollection 2019. PMID 31908502
- [Background] Meng L, Pourali S, Hitchcock MM, Ha DR, Mui E, Alegria W, Fox E, Diep C, Swayngim R, Chang A, Banaei N, Deresinski S, Holubar M. Discontinuation Patterns and Cost Avoidance of a Pharmacist-Driven Methicillin-Resistant Staphylococcus aureus Nasal Polymerase Chain Reaction Testing Protocol for De-escalation of Empiric Vancomycin for Suspected Pneumonia. Open Forum Infect Dis. 2021 Mar 4;8(4):ofab099. doi: 10.1093/ofid/ofab099. eCollection 2021 Apr. PMID 34386545
- [Derived] De Vita E, Segala FV, Cavallin F, Guido G, Frallonardo L, Cotugno S, Pellegrino C, Di Gennaro F, Saracino A. Rapid de-escalation of anti-MRSA therapy guided by S. aureus nares screening for patients with pneumonia: protocol of a randomized controlled trial (SNAP study). Front Med (Lausanne). 2024 Sep 10;11:1416904. doi: 10.3389/fmed.2024.1416904. eCollection 2024. PMID 39318595
- See also: Antimicrobial resistance surveillance in Europe - 2023 — https://www.ecdc.europa.eu/en/publications-data/antimicrobial-resistance-surveillance-europe-2023
- See also: Rapporto AR-ISS - I dati 2022 - Istituto Superiore di Sanità — https://www.epicentro.iss.it/antibiotico-resistenza/ar-iss-rapporto